CLINICAL TRIAL: NCT05157048
Title: Acute Effects of Cigarette Packaging and Charcoal Filtration on Perceptions, Use Behaviors, and Harm Exposure
Acronym: SKY Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Andrew Strasser, Research Professor of Psychiatry, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: UPCC 05021; IRB 849152 (Other: Penn CTSRMC)
Record Dates: First submitted 2021-10-13; First posted 2021-12-14 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-08

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Single-session study utilizing a 2 x 2 mixed factorial design
Who Masked: Participant
Masking Description: Participants will be blinded to both the marketing and cigarette condition manipulations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Light pack color (Experimental): Participants will be randomized to one of two pack color conditions: light or dark. Those in the light pack color condition will be given Natural American Spirit Sky packs.
  Interventions: Other: Charcoal-filtered cigarette; Other: Non-charcoal filtered cigarette
- Dark pack color (Experimental): Participants will be randomized to one of two pack color conditions: light or dark. Those in the dark pack color condition will be given Natural American Spirit Black packs.
  Interventions: Other: Charcoal-filtered cigarette; Other: Non-charcoal filtered cigarette

INTERVENTIONS:
Other: Charcoal-filtered cigarette — Participants will smoke two visually identical cigarettes, one with a charcoal filter and one with a non-charcoal filter, in counterbalanced order. The charcoal filter cigarette will be a Natural American Spirit Sky cigarette; the non-charcoal filter cigarette will be a Natural American Spirit Orange cigarette.
  Other Names: Product
Other: Non-charcoal filtered cigarette — Participants will smoke two visually identical cigarettes, one with a charcoal filter and one with a non-charcoal filter, in counterbalanced order. The charcoal filter cigarette will be a Natural American Spirit Sky cigarette; the non-charcoal filter cigarette will be a Natural American Spirit Orange cigarette.
  Other Names: Product

SUMMARY:
This single laboratory session pilot study will examine the acute effects of cigarette filter type and packaging on initial product perceptions, use, and exposure. Forty adult daily smokers will be randomized to smoke two study-supplied commercially-available cigarettes interspersed by 45 minutes, completing pre- and post-cigarette carbon monoxide and questionnaire measures. We will use a 2 x 2 mixed factorial design to manipulate cigarette filter type (within-subject: charcoal vs. non-charcoal) and packaging (between-subject: light vs. dark).

DETAILED DESCRIPTION:
We will recruit 40 adult daily, non-menthol smokers to a single 2-hr laboratory study where they will smoke two study-provided [commercially available] cigarettes, each for a 10-min ad lib period, and then complete product perception and use measures. Smoking sessions will be video recorded and scored to capture puffing behavior, and carbon monoxide (CO) assessments will be collected before and after smoking to assess changes in acute smoke exposure. We will use a 2 x 2 mixed factorial design to manipulate the study-provided cigarette's packaging (between subject factor: light colored 'Sky' package vs. black NAS package; both industry-made) and filter type (within-subject factor: charcoal filter vs. non-charcoal filter; cigarettes will appear identical despite differences in filter composition). Primary outcomes will be product perceptions (risk perceptions, subjective ratings), use behaviors (puffing behavior and purchase task), and acute toxicant exposure (changes in CO).

ELIGIBILITY:
Inclusion Criteria:

* Male and female smokers who are between 21 and 60 years of age and self-report smoking at least 5 cigarettes per day for at least the past 12 months.
* Smokers of primarily non-menthol cigarettes.
* Not currently undergoing smoking cessation treatment or trying to quit.
* Able to communicate fluently in English (speaking, writing, and reading).
* Capable of giving written informed consent.

Exclusion Criteria:

Subjects who self-report and/or present with the following criteria will not be eligible to participate in the study:

Smoking Behavior

1. Use of menthol cigarettes as preferred/regular brand (defined as using >20% of the time).
2. Use of research cigarettes in the past 6 months (i.e., past 6-month participation in applicable previous CIRNA studies).
3. Enrollment or plans to enroll in a smoking cessation program in the next month.
4. Provide an initial Carbon Monoxide (CO) reading < 5 parts per million (ppm).

Alcohol/Drugs

1. History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse.
2. Current alcohol consumption that exceeds 25 standard drinks/week.

Medical

1. Women who are pregnant, planning a pregnancy, and/or lactating.
2. Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the completion of procedures included within this protocol. Notable impairments will be evaluated by the PI and eligibility will be determined on a case-by-case basis.
3. Color blindness.
4. Serious or unstable disease within the past 12 months (e.g. heart disease, cancer). Applicable conditions will be evaluated by the Principal Investigator and eligibility will be determined on a case-by-case basis.

Psychiatric

As determined by self-report:

1. Lifetime history or current diagnosis of psychosis, bipolar disorder, and/or schizophrenia.
2. Current diagnosis of major depression. Subjects with a history of major depression, in remission for 6 months or longer, are considered eligible.

Other

Additionally, participants may be deemed ineligible for any of the following general reasons at any point throughout the study, as well as during the initial telephone screen, at the discretion of the PI:

* Significant non-compliance with protocol and/or study design.
* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact study data.
* Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited individuals from the greater Philadelphia area from March 2022 through February 2023 using print and digital media advertisements and through contacting previous participants and individuals registered with an institutional clinical research database.
Pre-assignment Details: Of the 42 individuals who signed the consent form and enrolled in the study, 2 did not meet post-enrollment inclusion criteria, resulting in 40 participants being randomized to study conditions / completing the single session.
  To clarify our mixed design, all subjects sampled each filter type, but half of the sample received cigarettes in a black pack and half received cigarettes in light packs. Thus there are 2 groups, not 4, for which we present participant flow and sample characteristics.
Groups:
- Light Pack Color: All participants smoked two visually identical cigarettes, one with a charcoal filter and one with a non-charcoal filter (within-subject factor), in counterbalanced order. Participants were randomized to receive study cigarettes in one of two pack color conditions: light or dark (between-subject factor). Those in the light pack condition received cigarettes in Natural American Spirit Sky packs.
- Dark Pack Color: All participants smoked two visually identical cigarettes, one with a charcoal filter and one with a non-charcoal filter (within-subject factor), in counterbalanced order. Participants were randomized to receive study cigarettes in one of two pack color conditions: light or dark (between-subject factor). Those in the dark pack condition received cigarettes in Natural American Spirit Black packs.
Period: Overall Study
Arm/Group | Light Pack Color | Dark Pack Color
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Light Pack Color; Dark Pack Color: All participants will be smoke two visually identical cigarettes, one with a charcoal filter and one with a non-charcoal filter (within-subject conditions), in counterbalanced order. Participants will be randomized to receive study cigarettes in one of two pack color conditions: light or dark (between-subject factor).
- Total: Total of all reporting groups
Arm/Group | Light Pack Color | Dark Pack Color | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (10.7) | 45.0 (13.0) | 46.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White vs. Other Categories: White | 16 | 14 | 30
  White vs. Other Categories: Non-White | 5 | 5 | 10
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Assessed using the question, "In the past 7 days, about how many cigarettes have you smoked per day?"
  cigarettes per day | 13.1 (4.4) | 15.6 (7.7) | 14.3 (6.2)
Years smoking regularly [Mean (Standard Deviation); unit: years] | 29.9 (11.4) | 27.7 (16.1) | 28.9 (13.7)
Nicotine dependence [Mean (Standard Deviation); unit: units on a scale] — Assessed using the Fagerstrom Test for Cigarette Dependence (FTCD), a 6-item, self-report measure of nicotine dependence. Items are summed to a score ranging from 0-10, with greater scores indicating greater nicotine dependence.
  units on a scale | 4.9 (1.7) | 5.0 (2.6) | 4.9 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Puffs Taken (Video-scored Smoking Behavior Outcome 1)
Description: Smoking behaviors were assessed using video-scored measures of smoking topography (i.e., puffing behavior), including number of puffs taken, total puffing duration, and total interpuff interval (time between puffs). Briefly, research staff used a digital timestamp feature in an open-source video editing software to estimate start and end times for individual puffs based on various physical cues (e.g., inhaling, glowing cigarette tip), prioritizing overall puffing behaviors (e.g., multiple occurrences of tip glowing without removing the cigarette from the mouth ["stutter puffs"] were treated as a single puff).
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: puffs
Groups:
- Light Pack Color; Dark Pack Color: All participants will smoke two visually identical cigarettes varying in filter type (within-subject condition: charcoal and non-charcoal filter), in counterbalanced order. Participants will be randomized to receive cigarettes in one of two pack colors (between-subject-condition: light or dark).
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
puffs
  Charcoal filtered cigarette | 15.8 (1.8) | 16.7 (1.9)
  Non-charcoal filtered cigarette | 19.1 (2.3) | 19.6 (2.4)

2. Primary Outcome: Total Puffing Duration (Video-scored Smoking Behavior Outcome 2)
Description: as for outcome 1
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
seconds
  Charcoal filtered cigarette | 30.4 (4.3) | 32.6 (4.5)
  Non-charcoal filtered cigarette | 41.4 (6.1) | 41.2 (6.4)

3. Primary Outcome: Total Interpuff Interval (Video-scored Smoking Behavior Outcome 3)
Description: as for outcome 1
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
seconds
  Charcoal filtered cigarette | 257.7 (28.9) | 290.4 (30.3)
  Non-charcoal filtered cigarette | 267.9 (28.8) | 275.0 (30.3)

4. Primary Outcome: Correct Beliefs About Reduced Risks
Description: Risk beliefs were captured using an 8-item scale that asked participants to compare each study cigarette to 'regular' cigarettes on eight statements (i.e., "lower in nicotine", "lower in tar", "less addictive", "less likely to cause cancer", "has fewer chemicals", "is healthier", "makes smoking safer", "helps people quit smoking") using a 5-point response scale (1='definitely untrue', 5='definitely true'). Responses were scored dichotomously ("untrue" responses scored as correct; "unsure"/"true" responses scored as incorrect) and summed to create an overall beliefs measure. Thus, responses are possible on a scale of 0-8, with a score of 0 indicating no correct beliefs and 8 indicating the participant was correct on all belief items.
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal filtered cigarette | 3.8 (0.6) | 3.8 (0.6)
  Non-charcoal filtered cigarette | 2.9 (0.6) | 3.2 (0.6)

5. Primary Outcome: Perceived Health Risks Summary Score
Description: Perceived health risks were assessed using the mean of six items that asked participants to indicate on a 7-point Likert scale (1 = "very low risk", 7 = "very high risk") their risk of developing smoking-related health conditions (i.e., lung cancer, heart disease, stroke, emphysema, respiratory infections, and other cancers) from regular use of each study cigarette.
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal-filtered cigarette | 5.6 (0.3) | 5.4 (0.3)
  Non-charcoal filtered cigarette | 5.3 (0.3) | 5.3 (0.3)

6. Primary Outcome: Product Harshness (Subjective Rating Subscale 1)
Description: Subjective ratings were assessed with THE Cigarette Rating Scale, a 100 mm visual analog scale used by the tobacco industry and our laboratory to assess 14 characteristics; higher scores generally indicate more favorable ratings (e.g., taste: 0 = "bad," 100 = "good"). We examined mean scores from three subscales generated from these items to assess domains of product harshness, smoking satisfaction, and positive sensory experience. We also explored a fourth 'cleanliness' subscale created by averaging two exploratory items assessing "chemical vs. tobacco taste" and "dirty vs. clean body feeling" based on qualitative data from a related pilot study. All subscale scores have a range of 0-100, with higher scores generally indicative of more favorable ratings.
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal filtered cigarette | 42.1 (4.4) | 42.6 (4.6)
  Non-charcoal filtered cigarette | 24.7 (4.7) | 26.2 (5.0)

7. Primary Outcome: Smoking Satisfaction (Subjective Rating Subscale 2)
Description: as for outcome 6
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal filtered cigarette | 65.8 (4.2) | 55.9 (4.4)
  Non-charcoal filtered cigarette | 43.0 (4.9) | 36.2 (5.2)

8. Primary Outcome: Positive Sensory Experience (Subjective Rating Subscale 3)
Description: as for outcome 6
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal filtered cigarette | 59.3 (5.2) | 47.5 (5.4)
  Non-charcoal filtered cigarette | 48.4 (5.2) | 48.1 (5.4)

9. Primary Outcome: Cleanliness (Subjective Rating Subscale 4)
Description: as for outcome 6
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
score on a scale
  Charcoal filtered cigarette | 72.4 (5.8) | 47.7 (6.1)
  Non-charcoal filtered cigarette | 70.5 (5.5) | 49.3 (5.8)

10. Primary Outcome: Carbon Monoxide (CO) Boost
Description: CO will be measured in parts per million (ppm) using the Vitalograph BreathCO carbon monoxide monitor (Lenexa, KS) at the onset of the laboratory visit, as well as before and after each cigarette smoked. CO boost - the change in CO values resulting from smoking a cigarette - crudely estimates smoke exposure due to smoking an individual cigarette.
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: parts per million
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
parts per million
  Charcoal-filtered cigarette | 4.6 (0.7) | 3.6 (0.7)
  Non-charcoal filtered cigarette | 5.0 (0.7) | 2.4 (0.7)

11. Secondary Outcome: Intensity
Description: A hypothetical cigarette purchase task, asked how many study cigarettes participants would purchase in a typical day across a range of escalating prices from free up to $1.45 per cigarette, chosen to reflect double the current median price of Natural American Spirit brands in the U.S. However, because 35-40% of participants failed to reach breakpoint (i.e., the price point at which consumption drops to 0), we report observed values for demand index of intensity (number of cigarettes consumed for free) only.
Time Frame: Session 1; assessed after smoking each of the two study cigarettes (i.e., after each filter condition)
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Light Pack Color | Dark Pack Color
Number analyzed (Participants) | 21 | 19
cigarettes per day
  Charcoal-filtered cigarette | 15.2 (2.5) | 19.7 (2.7)
  Non-charcoal filtered cigarette | 12.7 (2.5) | 18.8 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected as this study was comprised of a single session.
Description: Adverse event data were not collected as this study was comprised of a single session.
Arm/Group | Light Pack Color | Dark Pack Color
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This sample may not reflect the general smoking population or intended consumers of Sky; because we used commercial packages to examine their real-world marketing effects, we could not disentangle effects of color from other packaging elements; the low maximum price used in the purchase task limited the utility of this measure as an outcome; findings reflect reactions to charcoal-filtered cigarettes and their packaging after an acute, blinded one-time exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT05157048/Prot_SAP_000.pdf